CLINICAL TRIAL: NCT05150457
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BNA035 in Patients With Advanced Solid Tumors
Brief Title: Safety and Preliminary Efficacy of BNA035 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Binacea Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNA035-101
Record Dates: First submitted 2021-11-11; First posted 2021-12-09 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Refractory Solid Tumors
Keywords: Cancer; Advanced cancer; Recurrent cancer; Solid tumor; Metastatic cancer; Refractory cancer
MeSH Terms: conditions — Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Phase, Dose Level 1 (Experimental): Starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles.
  Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035
- Dose Escalation Phase, Dose Level 2 (Experimental): 3 times the starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035
- Dose Escalation Phase, Dose Level 3 (Experimental): 10 times the starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035
- Dose Escalation Phase, Dose Level 4 (Experimental): 30 times the starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035
- Dose Escalation Phase, Dose Level 5 (Experimental): 100 times the starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035
- Dose Escalation Phase, Dose Level 6 (Experimental): 200 times the starting dose level of BNA035 administered as an IV infusion once weekly in 28 day cycles Drug: BNA035 Administered once weekly as an IV infusion at the assigned dose level in 28 day cycles
  Interventions: Drug: BNA035

INTERVENTIONS:
Drug: BNA035 — Anti-epidermal growth factor receptor (Anti-EGFR) and anti-cluster of differentiation 137 (anti-CD137) bispecific antibody

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of BNA035 in order to determine the maximum tolerated dose (MTD) and Recommended Phase 2 dose (RP2D) and to evaluate the preliminary efficacy for each combination regimen.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment in this study:

1. Male or female ≥ 18 years of age.
2. Histologically or cytologically confirmed advanced malignant solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
3. Measurable disease as per RECIST 1.1, or per Response Assessment in Neuro-Oncology (RANO) criteria for patients with glioblastoma multiforme and documented by computed tomography (CT) and/or magnetic resonance imaging (MRI).
4. All persisting toxic effects of any prior anti-tumor therapy resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 Grade ≤ 1 or baseline before the first dose of study drug (with the exception of alopecia [Grade 1 or 2 permitted] and neurotoxicity [Grade 1 or 2 permitted]).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
6. Life expectancy of ≥ 3 months, in the opinion of the Investigator.
7. Adequate organ function defined as follows:

   1. Hematologic: Platelets ≥ 100 x 109/L; Hemoglobin ≥ 9.0 g/dL; Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (without blood transfusion, platelet transfusion, or growth factors within previous 7 days of the hematologic laboratory values obtained at Screening visit).
   2. Hepatic: Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≤ 5 x ULN); Total or conjugated bilirubin ≤ 1.5 x ULN.
   3. Renal: Creatinine clearance (CLcr) ≥ 45 mL/min as calculated by the Cockcroft Gault method.
8. Coagulation: Patients on full-dose oral anticoagulation, except warfarin, which is an excluded medication, must be on a stable dose (minimum duration 14 days). Patients on low molecular weight heparin will be allowed.
9. Negative serum pregnancy test for female patients.
10. If of childbearing potential, female patients must be willing to use highly effective double contraceptive measures starting with the Screening visit through 90 days after the last dose of study treatment.

    Double contraception is defined as a condom AND one other form of the following:
    * Established hormonal contraception (with approved oral contraceptive pills, long-acting implantable hormones, injectable hormones);
    * A vaginal ring or an intrauterine device (IUD);
    * Documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner).

    Women not of childbearing potential must be post-menopausal for ≥ 12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.

    Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not considered highly effective methods of birth control. Complete abstinence for the duration of the study through 90 days after the last dose of study treatment is acceptable if this is the established and preferred contraception for the patient.

    Female patients who are in same-sex relationships are not required to use contraception.
11. Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the Screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    Acceptable methods of contraception include:
    * Vasectomy (> 30 days since vasectomy with no viable sperm);
    * Surgical sterility in female partner(s) (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy);
    * Double contraception, condom AND the use of an effective contraceptive for the female partner that includes: oral contraceptive pills, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD.

    Patients with same-sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.

    Note: Abstinence is acceptable if this is the established and preferred contraception method for the patient.
12. Males must not donate sperm for at least 90 days after the last dose of study drug.
13. Able and willing to provide written informed consent to participate in the study.
14. Patients with history of human immunodeficiency virus (HIV) infection should have a cluster of differentiation 4+ (CD4+) T cell count ≥ 350 cells/µL at Screening.
15. Patients with serological evidence of chronic hepatitis B virus infection (HBV) should have HBV viral load below the limit of quantification at Screening.
16. Patients with serological evidence of hepatitis C virus infection (HCV) should have completed curative antiviral treatment and have HCV viral load below the limit of quantification at Screening.
17. Patients must not be using immunosuppressive medication > 10 mg prednisolone per day or equivalent, or 2 mg dexamethasone for glioblastoma multiforme (GBM) patients, within 14 days prior to the first dose of the study drug. Note: Use of immunosuppressive medications as prophylaxis in patients with contrast allergies are acceptable. In addition, temporary uses of corticosteroids considered non-clinically significant may be approved on a case-by-case basis in discussion with the Sponsor.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from this study:

1. Pregnant or lactating or planning to become pregnant (self or partner) at any time during the study, including the Follow-up Period.
2. History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the Investigator or Medical Monitor, would pose a risk to patient safety or interfere with the study evaluations, procedures, or completion.
3. History of ≥ Grade 3 AEs during prior treatment with an immune checkpoint inhibitor, or history of discontinuation of treatment with an immune checkpoint inhibitor due to AEs. Previous Grade 3 immune-related adverse events (irAEs) if not considered by the Investigator to increase the patient's risk for investigational product (IP) related AEs, may be approved on a case-by-case basis in discussion with the Sponsor (e.g., hypothyroidism on stable thyroxine replacement, adrenal insufficiency on stable hormone replacement therapy, diabetes on stable insulin therapy).
4. Active or history of prior autoimmune disease with the exception of:

   * Hashimoto's Thyroiditis on stable thyroid replacement therapy;
   * Type 1 Diabetes Mellitus (T1DM) on stable insulin therapy;
   * Other prior autoimmune disorders not considered to put at higher risk for irAEs, based on Investigator judgment and approved by the Sponsor on a case-by-case basis (e.g., rheumatoid arthritis).

   The use of stable and controlled low dose steroids is acceptable.
5. Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases, and if taking corticosteroids, are on stable or decreasing doses for at least 7 days from first dose of study drug. Patients with GBM are eligible, if meeting all other inclusion criteria and no exclusion criteria.
6. Patients with hepatocellular carcinoma are excluded.
7. Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection requiring systemic therapy, active or chronic bleeding event within 28 days prior to first dose of study drug, or psychiatric illness/social situation that would limit compliance with study requirements as judged by the treating physician.
8. Current or previous interstitial lung disease.
9. Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, serious uncontrolled cardiac arrhythmia, cerebral vascular accident, coronary/peripheral artery bypass graft surgery, or pulmonary embolism within the last 6 months of first dose of study drug. Patients with small pulmonary embolism not thought to put patients at higher risks of AEs may be allowed on a case-by-case basis in discussion with the Sponsor.
10. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days of the first dose of study drug.
11. Symptomatic with uncontrolled ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions (including thoracentesis or paracentesis), with no need for repeating paracentesis/thoracentesis within 7 days prior to Cycle 1 Day 1 (C1D1), is eligible.
12. Minor surgical procedure(s) within 7 days of enrollment, or not yet recovered from prior surgery (placement of central venous access device, fine needle aspiration, or endoscopic biliary stent ≥ 1 day before enrollment is acceptable).
13. Prior systemic radiation therapy completed within 4 weeks of the first dose of study drug, prior local radiation therapy completed within 2 weeks of C1D1, or radiopharmaceuticals (strontium, samarium) within 8 weeks of C1D1. Palliative radiotherapy given within 14 days prior to the first dose of study drug may be approved on a case-by-case basis in discussion with the Sponsor.
14. Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy) within 28 days or 5 half-lives, whichever is shorter, of study drug dosing (6 weeks for nitrosoureas, mitomycin C, or molecular agents with t1/2 > 10 days).
15. History of long QT syndrome or additional risk factors for Torsades de Pointes or whose corrected QT interval (QTc) measured (Fridericia method) at Screening is prolonged (> 480 ms).
16. Use of concomitant medications that prolong QT/QTc interval at Screening that cannot be discontinued.
17. Known hypersensitivity to study drug, the metabolites or formulation excipients.
18. Use of any prohibited concomitant medications as described in Section 5.7.3 and any investigational agent within 2 weeks of study treatment initiation.
19. Received live virus vaccination within 30 days of first dose of study treatment. Seasonal flu vaccines that do not contain live virus are permitted.
20. History of hematologic stem cell transplant or solid organ transplant.
21. Participation or plans to participate in another interventional clinical study while taking part in this protocol; participation in an observational study is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Determination of the Maximum Tolerated Dose (MTD) Recommended Phase 2 Dose (RP2D) of BNA035 in patients with advanced solid tumors. | From first dose of BNA035 (Cycle 1 Day 1) through the end of the DLT period (28 days from Cycle 1 Day 1)
  Evaluated by the number of dose-limiting toxicities (DLT) graded using NCI CTCAE v 5.0
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From first dose of BNA035 through 90 days after the last BNA035 dose)
  To examine the incidence of clinical and laboratory adverse events after multiple doses of BNA035 in the dose escalation and dose expansion phases.

SECONDARY OUTCOMES:
Peak Plasma Concentration of BNA035 | Days 1, 2, 3, 5, and 8 of Cycle 1 and 2; Day 15 of Cycle 1; Day 1 of Cycles 3, 4, and 5 (each cycle is 28 days); after last BNA035 treatment (up to 1 year)
  To evaluate the maximum observed concentration (Cmax) after single and repeated IV weekly doses of BNA035
Area under the plasma concentration of BNA035 | Days 1, 2, 3, 5, and 8 of Cycle 1 and 2; Day 15 of Cycle 1; Day 1 of Cycles 3, 4, and 5 (each cycle is 28 days); after last BNA035 treatment (up to 1 year)
  To evaluate the area under the curve (AUC) plasma-concentration after single and repeated IV weekly doses of BNA035
Half-life of BNA035 | Days 1, 2, 3, 5, and 8 of Cycle 1 and 2; Day 15 of Cycle 1; Day 1 of Cycles 3, 4, and 5 (each cycle is 28 days); after last BNA035 treatment (up to 1 year)
  To evaluate the half-life of BNA035 after single and repeated IV weekly doses
Investigate immunogenicity of BNA035 | Day 1 of Cycle 1; Day 1 of every other Cycle thereafter (each cycle is 28 days); after last BNA035 treatment (up to 1 year)
  Evaluated by the incidence and characteristics of anti-drug antibody (ADA) of BNA035

CONTACTS AND LOCATIONS:
Overall Officials: Josh Xiao, PhD, Study Chair — Binacea Pharma, Inc.
Locations (3):
- Australia (3):
  - St George Private Hospital, Kogarah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - St. Vincents Hospital Melbourne, Fitzroy, Victoria